CLINICAL TRIAL: NCT03829059
Title: Retrospective Clinico-pathological Examinations on Different Histological/ Immunohistological and Molecularpathological Types of Epulides and Central Giant Cell Lesions of the Jaws
Brief Title: Histological/ Immunohistological and Molecularpathological Types of Epulides and Central Giant Cell Lesions of the Jaws
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: GCG
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Epulis
MeSH Terms: conditions — Gingival Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective study will evaluate the patient collective of the Division of Oral Surgery and Orthodontics, Department of Dental Medicine and Oral Health and of the Division of Cranio-Maxillofacial Surgery at the Medical University Graz concerning the frequency of epulis/giant cell lesion or underlying differential diagnoses and immunophenotypes as well as the resulting treatment methods and their success and compare these with international results

DETAILED DESCRIPTION:
Different histopathological differential diagnoses can underlay the clinical presentation of an epulis. Often the immunophenotype of these lesions is of particular importance. This also holds for the the central giant cell lesion.

This study will evaluate the patient collective of the Division of Oral Surgery and Orthodontics, Department of Dental Medicine and Oral Health and of the Division of Cranio-Maxillofacial Surgery at the Medical University Graz concerning the frequency of epulis/giant cell lesion or underlying differential diagnoses and immunophenotypes as well as the resulting treatment methods and their success and compare these with international results.

This is a retrospective study using electronic patient records, written records, operative reports of the Division of Oral Surgery and Orthodontics, Department of Dental Medicine and Oral Health and of the Division of Cranio-Maxillofacial Surgery at the Medical University Graz in the period from 1986 to March 2018. It is intended to gather the data within 12 months and analyze statistically subsequently.

ELIGIBILITY:
Inclusion Criteria:

* existence of a medical history and a histopathological finding of the surgical specimen
* patients treated in the outpatient clinic for diseases of oral mucosa of the Division of Oral Surgery and Orthodontics, Department of Dental Medicine and Oral Health and of the Division of Cranio-Maxillofacial Surgery at the Medical University Graz between 1986 and March 2018

Exclusion Criteria:

* absence of a medical history or a histopathological finding.

Ages: 7 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patient cohort comprises 101 patients treated in the outpatient clinic for diseases of oral mucosa of the Division of Oral Surgery and Orthodontics, Department of Dental Medicine and Oral Health and of the Division of Cranio-Maxillofacial Surgery at the Medical University Graz in the period from 1986 to March 2018.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Frequency of histological pathological differential diagnoses. | time period of evaluation from 1986 to March 2018
Frequency of immunohistochemical pathological differential diagnoses. | time period: from 1986 to March 2018
Frequency of molecular pathological differential diagnoses. | time period from 1986 to March 2018

SECONDARY OUTCOMES:
Frequency of recurrences | time period from 1986 to March 2018
  depending on differential diagnoses and therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University, Graz, Austria